CLINICAL TRIAL: NCT01442207
Title: Cerclage Placement for the Prevention of Preterm Birth in Women With Placenta Previa - A Multicenter Randomized Controlled Trial
Brief Title: Cerclage for Prevention on Preterm Birth in Women With Placenta Previa
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of randomized participants
Sponsor: Obstetrix Medical Group (Industry)
Responsible Party: Sponsor
Organization: Pediatrix (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OBX 0018
Record Dates: First submitted 2011-09-15; First posted 2011-09-28 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Premature Birth; Placenta Previa
Keywords: Premature Birth; Placenta Previa
MeSH Terms: conditions — Premature Birth; Placenta Previa | interventions — Cerclage, Cervical; Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placement of Cervical Cerclage (Active Comparator): Cervical Cerclage is to be placed in an inpatient hospital setting within 24 to 72 hours of being assigned to this treatment group
  Interventions: Procedure: Placement of a Cervical Cerclage
- Expectant Management (Placebo Comparator): Participants assigned to the expectant management group will be followed by their doctor and managed per standard management which includes:
  * Standard management for placenta previa.
  * Hospital admission for vaginal bleeding/hemorrhage
  * Antenatal corticosteroids > 24w0d of gestation
  * Tocolytic therapy per physician's discretion
  * Magnesium sulfate for neuroprotection
  * Fetal Heart Rate Monitoring
  * Avoidance of digital examinations of the cervix
  * Elective delivery no earlier than 36w0d gestation unless indicated (uncontrolled hemorrhage, imminent delivery, Premature rupture of the membranes (PROM) > 34 wks, worsening maternal or fetal condition )
  * Fetal Fibronectin (fFN) test collected at the time of transvaginal Ultrasound.
  Interventions: Procedure: Standard Expectant Management

INTERVENTIONS:
Procedure: Placement of a Cervical Cerclage — Surgical placement of a cervical cerclage
  Other Names: cerclage
  Arms: Placement of Cervical Cerclage
Procedure: Standard Expectant Management — Participants assigned to the expectant management group will be followed by their doctor and managed per standard management which includes:
  * Standard management for placenta previa.
  * Hospital admission for vaginal bleeding/hemorrhage
  * Antenatal corticosteroids > 24w0d of gestation
  * Tocolytic therapy per physician's discretion
  * Magnesium sulfate for neuroprotection
  * Fetal Heart Rate Monitoring
  * Avoidance of digital examinations of the cervix
  * Elective delivery no earlier than 36w0d gestation unless indicated (uncontrolled hemorrhage, imminent delivery, PROM > 34 wks, worsening maternal or fetal condition )
  * Fetal Fibronectin (fFN) test collected at the time of transvaginal Ultrasound.
  Other Names: Expectant Management
  Arms: Expectant Management

SUMMARY:
The purpose of the study is to compare the role of cervical cerclage versus expectant management in women with complete placenta previa (≥ 10mm over internal os) presenting with shortened cervical length ( ≥ 10mm and ≤ 30mm) between 18w0d and 26w0d of pregnancy.

DETAILED DESCRIPTION:
The purpose of this study is to perform a large multi-center randomized trial comparing the role of cervical cerclage versus expectant management in women with placenta previa presenting with shortened cervical length ( ≥ 10mm and ≤ 30mm) between 18w0d and 26w0d of gestation. In addition, the role of fetal fibronectin (fFN) for the prediction of preterm birth and hemorrhage will be elucidated. The hypothesis is that placement of a cervical cerclage between 18w0d to 26w0d in patients with a short cervix and complete placenta previa will decrease preterm birth as compared to expectantly managing these patients.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy, ≥ 18yrs old
* GA 18w0d to 26w0d inclusive @ time of enrollment
* Documentation of complete placenta previa (≥ 10mm over internal os)
* Agrees to participate in trial and signs/date an informed consent form.

Exclusion Criteria:

* Contraindication to expectant management (i.e. active labor, Non-reassuring fetal heart rate (NRFHR), Intrauterine fetal demise (IUFD), uncontrolled hemorrhage)
* Fetal condition likely to cause serious neonatal morbidity independent of GA (e.g. hydrops, fetal viral infections, fetal malformations likely to need surgery like hydrocephalus, neural tube defects, cardiac defects, abdominal wall defects)
* Known uterine anomaly at time of enrollment
* History of two or more prior cesarean deliveries
* Suspected placenta accrete, increta or percreta on US at enrollment
* Cervical cerclage present at time of enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Gestational age (GA) at birth | measure taken in the first 23 hours after birth.
  The gestational age (GA) of the baby noted at birth

SECONDARY OUTCOMES:
Newborn Birth weight | measured within 1-2 days after birth
  Newborn Birth weight measure within 1-2 days after birth.
Need for Maternal Blood Product replacement | measured from the time participant is enrolled in the study until 30 days after delivery.(approximately 40 weeks)
  Maternal need for blood product replacement such as Fresh Frozen Plasma.
Number of participants delivering prematurely following hemorrhage who have a positive fFN test. | measured at delivery
  Measure the total number of patients (participants) who delivered prematurely as a result of hemorrhage who also had a positive fFN test.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Stafford, MD, Principal Investigator — Obstetrix Medical Group of Tucson.